CLINICAL TRIAL: NCT06431542
Title: Comparison of the Efficacy of Patient Self-Application Versus Physician Application of Triamcinolone Acetonide Econazole Cream in the Treatment of Otomycosis
Brief Title: Efficacy of Self Vs. Physician Application of Triamcinolone-Econazole in Otomycosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMZSYYKY2024-047
Record Dates: First submitted 2024-05-18; First posted 2024-05-28 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Otomycosis
Keywords: triamcinolone acetonide econazole cream; otomycosis
MeSH Terms: conditions — Otomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patient-applied medication group (Active Comparator): The doctor provided detailed instructions for the patient to self-apply Triamcinolone Acetonide Econazole Cream to the external auditory canal once daily for two weeks.
  Interventions: Procedure: patient-applied Triamcinolone Acetonide Econazole Cream
- physician-applied medication group (Experimental): The doctor applied Triamcinolone Acetonide Econazole Cream for patients once every 2 to 3 days, for a total of three applications.
  Interventions: Procedure: physician-applied Triamcinolone Acetonide Econazole Cream

INTERVENTIONS:
Procedure: physician-applied Triamcinolone Acetonide Econazole Cream — The doctor applies the Triamcinolone Acetonide Econazole Cream onto a thin cotton swab and gently inserts it deep into the ear canal, evenly spreading the cream around the sides of the ear canal and on the surface of the eardrum.
  Arms: physician-applied medication group
Procedure: patient-applied Triamcinolone Acetonide Econazole Cream — The patient applies Triamcinolone Acetonide Econazole Cream in the external auditory canal at home using a cotton swab.
  Arms: patient-applied medication group

SUMMARY:
to analyze the clinical characteristics, types of Fungal Infections, and comparison of the efficacy of patient self-application versus physician application of triamcinolone acetonide econazole cream in otomycosis treatment.

DETAILED DESCRIPTION:
The study analyzes the clinical characteristics, including symptoms and physical examinations, as well as the types of fungal infections. It compares the efficacy of patient self-application versus physician application of triamcinolone acetonide econazole cream in treating otomycosis two weeks after starting treatment. Furthermore, the study also compares the recurrence rates six months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.The chief complaint was ear discomfort, including tinnitus, a feeling of blockage or fullness, pruritis, otalgia, otorrhea and decreased hearing; 2. Physical examination findings:presence of fungal hyphae or accumulations that appear creamy or cheese-like or resembling abnormal earwax (crusts, films) , skin redness, erosion, swelling, or granulation tissue within the ear canal; 3. Positive results in fungal culture.

Exclusion Criteria:

* The exclusion criteria included otitis media, tympanic membrane perforation, and conditions post-radiotherapy.

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
treatment efficacy | 2 weeks
  Treatment efficacy is defined as the proportion of patients who are effective after two weeks of treatment. Effectiveness is defined by the absence of abnormalities in the external auditory canal and the alleviation of symptoms.

SECONDARY OUTCOMES:
recurrece rate | 3 months
  Recurrence rate is assessed three months later during a follow-up examination, where the presence of abnormal secretions in the ear canal and the recurrence of symptoms are noted.

CONTACTS AND LOCATIONS:
Overall Officials: Chunsheng Chunsheng, Principal Investigator — Xiamen University Zhongshan Hospital
Locations (1):
- Xiamen University Zhongshan Hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available within six months after the completion of the study and will remain accessible for at least ten years.
Access Criteria: The data will be open to peer-reviewed researchers. Researchers requesting access to the data must submit a research proposal and pass our review process. All data requestors must also adhere to a data use agreement.
URL: http://www.medresman.org